CLINICAL TRIAL: NCT05725837
Title: Effects of Paroxetine on Cardiovascular Function in Septic Patients: a Randomized Placebo Controlled Trial
Brief Title: Effects of Paroxetine on Cardiovascular Function in Septic Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude (Other)
Responsible Party: Principal Investigator, Felipe Dal Pizzol, Professor, Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Paroxetine
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Septic Shock; Sepsis
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Paroxetine

STUDY DESIGN:
Intervention Model Description: After 20 patients randomized the advisory board will unblind subjects to determine if the fluoxetine arm should be continued. Since it is not expected to have any beneficial effect of this treatment (it is only a comparative control to the effect of paroxetine on serotonin metabolism). Based on the decision of the committee the study could exclude the serotonin arm and the definitive sample size is going to be calculated.
  The fluoxetine group was removed from the study after analysis of the first 20 patients (as foreseen in the initial protocol, after 20 patients included the blind would be broken to determine the final sample size) as it did not present an apparent benefit in the primary outcome. Considering that it had been included as a comparator for the effect of paroxetine on serotonin metabolism, and no beneficial effect from its use was anticipated, the study management committee decided to withdraw it.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 40mg, single dose a day, by mouth or enteric tube
  Interventions: Drug: Paroxetine
- Paroxetine (Experimental): 40mg, single dose a day, by mouth or enteric tube
  Interventions: Drug: Paroxetine

INTERVENTIONS:
Drug: Paroxetine — Paroxetine, 40mg/day, once a day, for 05 consecutive days or 24 hours after shock resolution

SUMMARY:
It is known that septic shock is characterized by arterial hypotension, decreased peripheral vascular resistance and hyporeactivity to vasoconstrictor agents, with NO being an important mediator of this organ dysfunction. Data in the literature have shown that hyporeactivity to catecholamines is associated with a decrease in the density of α and ß receptors in the aorta and heart, respectively, as well as an increase in GRK2 levels and that NO contributes to the increase of this kinase in sepsis .

Based on this, it is hypothesized that cardiac dysfunction and decreased peripheral vascular resistance observed in sepsis may result from an increase in GRK2 activity and/or expression and its inhibition may be a relevant therapeutic target in septic shock patients. Based on this line, a measurable clinical benefit of paroxetine through the regulation of GRK2 expression in patients with septic shock is postulated.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age;
* Patient diagnosed with septic shock for less than 48 hours and using a minimum dose of noradrenaline (0.01 mcg/kg/min);
* Patients and/or legal guardians who consented to participate in the study through the free and informed consent term before randomization.

Exclusion Criteria:

* Pregnant women;
* Patients with inability to use the gastrointestinal tract;
* Patients with known intolerance to paroxetine and/or fluoxetine;
* Patients on concomitant use of medications that may potentiate the occurrence of serotonin syndrome (tramadol, citalopram, escitalopram, sertraline, desvenlafaxine, venlafaxine, duloxetine, sibutramine, bupropion, amitriptyline, nortriptyline, lithium);
* Patients in end-of-life care or with an expected survival of less than 24 hours at the time of eligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Time to vasopressor discontinuation | 28 days of enrollment
  Discontinuation of all vasopressors for at least 48 consecutive hours

SECONDARY OUTCOMES:
Cumulative vasopressor dose in the first 48 hours after randomization Translation results Cumulative vasopressor dose in the first 48 hours after randomization | 48 hours
  Dose of infused norephineprine and/or vasopressin during the first 48 hours after randomization
Variation in cardiovascular sequential organ failure assessment score score 24 to 120 hours after randomization | 120 hours
  Variation of the cardiovascular sequential organ failure assessment score score between baseline daily until 120 hours later. Cardiovascular sequential organ failure assessment score varies between 0 and +4 points, higher scores meaning worse cardiovascular dysfunction
Cumulative vasopressor dose for 120 hours after randomization | 120 hours
  Dose of infused norephineprine and/or vasopressin during 120 hours after randomization
Total sequential organ failure assessment score score variation 24 to 120 hours after randomization | 120 hours
  Variation of the total sequential organ failure assessment score score between baseline daily until 120 hours later. Total sequential organ failure assessment score varies between 0 and +24 points, higher scores meaning worse organ dysfunction
Length of stay in the ICU | 90 days
  time spent in ICU
Mortality during ICU stay | 90 daus
  Mortality in the ICU

OTHER OUTCOMES:
Neutrophilic levels of total and phosphorylated GRK2 | 120 hours
  Expression of GRK-2 measured by western blot in isolated neutrophils
Plasma levels of cytokines and chemokines | 120 hours
  Plasma levels of different cytokines and chemokines measured by ELISA
Internalization of CXCR2 receptors in neutrophils | 120 hours
  Internalization of receptors known to be influenced by GRK-2 inhibitor by flow cytometry

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Hospital Maternidade São José de Colatina, Colatina, Espírito Santo
  - Hospital São José, Criciúma, Santa Catarina

IPD SHARING:
Plan to Share IPD: Undecided